CLINICAL TRIAL: NCT04096885
Title: The Inselspital Surgical Cohort Study
Acronym: InSurg
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00576
Record Dates: First submitted 2019-08-30; First posted 2019-09-20 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Surgical Site Infection
Keywords: cohort; visceral surgery; biobank
MeSH Terms: conditions — Surgical Wound Infection | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Blood, urine and stool samples pre- and post-operative for microbiota, genomic and metabolomic analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- InSurg cohort: Patients who undergo elective or emergency surgery at the Department of Visceral Surgery and Medicine, Inselspital, Bern, who gave informed consent.
  Interventions: Diagnostic Test: Blood and urine samples, skin and stool swabs

INTERVENTIONS:
Diagnostic Test: Blood and urine samples, skin and stool swabs — Blood samples will be collected before surgery, on the first postoperative day and after 3-8 weeks. Urine samples will be collected after surgery and after 3-8 weeks. Stool and skin swabs will be collected before surgery.

SUMMARY:
Personalizing surgical care is of enormous clinical relevance, when considering the number of patients undergoing surgery in Switzerland every year. Currently, personalization is based on underlying or coexisting disease or alterations of laboratory values, but there is no accepted biological test available that may predict success or failure of surgery. Surgical site infections are the most common form of hospital-acquired infections. While the relevance of bacteria, antibiotics and intensive care support is well accepted, the impact of the individual host response remains poorly understood. The Investigators hypothesize that postoperative alterations of the metabolome allow identification of predictors of surgical complications in general, and surgical site infections in particular.

DETAILED DESCRIPTION:
The investigators will conduct a prospective cohort study aiming to identify the metabolic and genetic signature that is associated with surgical site infections. Secondary aims and outcomes include the influence of metabolome on response to anesthetic drugs and acute and chronic pain, surgery- and anesthesia-factors related to short- and long-term oncological outcome, metabolic response effect on infectious complications and rejection after transplantation, bacteria-specific immune responses to major surgery after 2-4 weeks after surgery, metabolomics and macrobiotic markers for postoperative ileus or anastomotic leakage, and the effect of the presence of multidrug resistant bacteria on surgical outcome. All patients undergoing surgery in the investigators' clinic and who gave informed consent will be included. A blood sample will be taken before surgery, on the first postoperative day and after 3-8 weeks. A Urine sample will be taken after surgery and after 3-8 weeks. Sink and rectal swabs will be acquired before surgery. The samples will be stored in a Biobank. Additionally, all data routinely captured during the treatment of the patient from the different data collection systems in use in the investigators' hospital will be coded and centralized in a single, cohort database

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery at the Department of Visceral Surgery and Medicine, Inselspital, University Hospital Bern
* Who gave General consent
* Study-specific written informed consent

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery at the Department of Visceral Surgery and Medicine, Inselspital, University Hospital Bern
Sampling Method: Non-Probability Sample
Enrollment: 1226 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of surgical site infection | 30 days
  Number of patients with surgical site infections 30 days postoperatively

SECONDARY OUTCOMES:
Stool - incidence of surgical site infections | 30 days
  Predictive value of preoperative stool sample for surgical site infections
Urine - incidence of surgical site infections | 30 days
  Predictive value of preoperative urine sample for surgical site infections
Blood - incidence of surgical site infections | 30 days
  Predictive value of pre and postoperative plasma metabolome for surgical site infections
Somatic genomic in surgical site infections | 30 days
  Predictive value of somatic genomic variations for surgical site infections
Informed Consent | 3 years
  Rate of inclusion for informed consenting
Biobanking | 3 years
  Rate of inclusion for full biobanking

OTHER OUTCOMES:
Intraoperative metabolomic Response to surgery | 8 weeks
  Metabolome will be extracted from the blood, skin, urine and stool samples analyzed using high resolution mass spectrometry. Metabolomic analysis will be obtained preoperatively in the outpatient setting (elective patients) or at the beginning (emergency patients) and end of the operation. Patterns of metabolites will be evaluated by untargeted analysis.
Disease-free survival after surgery | 3 years
  Disease-free survival after surgery in years will be recorded in oncological patients, and interpreted according to surgical and anesthesia-specific responses after abdominal surgery, in terms of metabolomics analysis of the blood, skin, urine and stool samples, as described above.
Recurrence-free survival after surgery | 3 years
  Recurrence-free survival after surgery in years will be recorded in oncological patients, and interpreted according to surgical and anesthesia-specific responses after abdominal surgery, in terms of metabolomics analysis of the blood, skin, urine and stool samples, as described above.
Overall survival after surgery | 3 years
  Overall survival after surgery in years will be recorded in oncological patients, and interpreted according to surgical and anesthesia-specific responses after abdominal surgery, in terms of metabolomics analysis of the blood, skin, urine and stool samples, as described above.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Beldi Guido, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No